CLINICAL TRIAL: NCT07084025
Title: Feasibility of Home-based Cognitive Strategy Training for Independence of Activities of Daily Living in Adults With Chronic Stroke
Brief Title: Home-based Cognitive Strategy Training for Daily Living in Adults With Chronic Stroke
Acronym: PRPP-HOME
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RC31/24/0579
Record Dates: First submitted 2025-07-16; First posted 2025-07-24 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Stroke; Cerebrovascular Disorders
Keywords: Cognitive strategy training; Task-based; Ecological; Performance; Activities of Daily Living
MeSH Terms: conditions — Stroke; Cerebrovascular Disorders

STUDY DESIGN:
Intervention Model Description: SCED (single-case design) in multiple baselines across 9 adults living at home with post-stroke cognitive disorders in chronic phase.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Perceive, Recall, Plan and Perform-Intervention (PRPP-I) (Experimental): task-based cognitive strategy training during activities appropriate for delivery in home-based setting.
  Interventions: Other: Perceive, Recall, Plan and Perform-Intervention protocol (PRPP-I)

INTERVENTIONS:
Other: Perceive, Recall, Plan and Perform-Intervention protocol (PRPP-I) — delivered over a 4-week period, in 12 sessions (45/60 min, 3 days a week for 4 weeks) for all patients according to the PRPP-I protocol. The intervention will be carried out by a PRPP-certified occupational therapist working on a Master's degree.
  It will consist of :
  * Implementation of training in functional cognitive strategies and meta-prompts through performance in home activities,
  * Repeated measurement of performance judgment criteria ;
  * Assessment of cognitive strategies
  * personalized implementation of the PRPP-I cognitive strategy training protocol.
  * Collection of feasibility modalities when tracking the intervention (e.g., time, transport, etc.).

SUMMARY:
This pilot experimental study aims to describe the feasibility of a cognitive strategy training protocol : PRPP-I, in activities of daily life across home-based setting for adults with chronic stroke for improvement of independence and quality of life. Aditionnally to examine preliminary effectiveness of PRPP-I protocol within a home-based setting on functional cognitive strategies, independence, quality of life and career burden.

DETAILED DESCRIPTION:
Stroke is the first cause of acquired disability in France causing impairments on independence. Depending on the area damaged, the impairments may vary. Indeed, these disorders can lead to a loss of autonomy and have an impact on independence in daily life activities. Following a stroke, most of patients retain long term consequences. 39 % of patients report cognitive impairment within three years after stroke. The prevalence of a cognitive impairment at 3 months post-stroke is estimated to be between 23 and 55 % impacting participation in daily life and quality of life. Due to reduced autonomy and participation restrictions, stoke patients need human assistance. It's estimated that 8,3 million people regularly provide home care to a dependent family member. Career time has demonstrated to increase with the level of dependency highlighting importance of rehabilitation of cognitive disorders after stroke for independence and caregiver burden prevention. Cognitive training during real-life activities warrants additional interest for improvement of autonomy in adults with stroke. Yet, majority of training is limited to hospital-based settings.

Perceive, Recall, Plan and Perform-Intervention protocol (PRPP-I) is aimed at delivering task-based cognitive strategy training during activities appropriate for delivery in home-based setting. The objective of this pilot study is to evaluate feasibility and preliminary effectiveness of the protocol of cognitive task-based strategy training on performance, independence and quality of life in adults with stroke within a home-based setting with a non-concurrent multiple baseline design.

Patients will be followed during 12 weeks over 3 phases. Phase A corresponds to the baseline, during this phase, there is no cognitive intervention. Intervention takes place during phase B. Patients will receive 3 sessions per week, lasting between 45 to 60 min during 4 weeks. PRPP-Intervention aimed at training cognitive strategies in an activity of daily living will be delivered. Subsequently, there will be a follow-up phase, during this period, patients will not have intervention. Assessments will be proposed to evaluate the possible results of the PRPP-Intervention.

ELIGIBILITY:
Patient's Main Eligibility criteria:

* Adult over 18 years of age;
* cognitive deficits (or Acquired Brain Injury) diagnosed due to ischemic or hemorrhagic, hemispheric or brainstem stroke, confirmed by brain imaging longer than 6 months;
* Patient with mild (<26/30 or <25/30 for patients aged 71-85 yr) or moderate ([18-25]/30) cognitive impairment, measured by the Montreal Cognitive Assessment test ;
* adults living in a home or community-based setting;
* Patient with a non-professional caregiver;

Patient's Main Exclusion criteria

* Neurological pathology other than stroke or psychiatric disorder;
* Significant cognitive impairment, according to MoCA score <18/30;
* Patient with severe aphasia, Boston Diagnostic Aphasia Examination score >2

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasability | From enrollment to the end of intervention at 4 weeks
  Composite outcome examine (1) the recruitment, (2) adherence to the protocol, (3) the implementation of the procedures (delivery) of the intervention and (4) the fidelity to intervention.
  (1) the adequate recruitment rate will be 9 participants who meet the inclusion criteria, assessed at 24 months; (2) Adherence will be adequate if > 80% of participants complete the PRPP-I protocol at home (≥80% of sessions) for 4 weeks, assessed at 4 weeks post-intervention; (3) Intervention procedures (delivery) will be assessed based on the implementation of resources for 12 PRPP-I intervention sessions delivered at home over 4 weeks, assessed at 4 weeks post-intervention; (4) Intervention fidelity, according to the PRPP-I protocol (i.e., intervention implementation) will be assessed using a standardized checklist. A procedural fidelity of ≥ 80% will be interpreted as adequate, calculated using the Tate & Perdices formula of 2019 and in accordance with SCRIBE guidelines.

SECONDARY OUTCOMES:
Functional Independence Measure (FIM) | At enrollment, Start of intervention (between 1 and 5 weeks post enrollment), End of intervention (between 5 and 9 weeks post enrollment), and 3-month follow-up post end of intervention
  The Functional Independence Measure (FIM) is used to assess the level of independence in activities of daily living in adults after stroke. It includes 18 items rated on a 7-point scale, where 1 indicates total assistance and 7 indicates complete independence. Thirteen items assess motor function (such as self-care and mobility), and five items assess cognitive function (such as communication and social interaction).
  The total score ranges from 18 (complete dependence) to 126 (complete independence). Motor and cognitive subscores can also be calculated, with maximum scores of 91 and 35 respectively.
  The FIM demonstrates good reliability, internal consistency, construct validity, and sensitivity to change. It is commonly used in clinical rehabilitation settings and aligns with current national and international guidelines for post-stroke functional assessment.

IPD SHARING:
Plan to Share IPD: No